CLINICAL TRIAL: NCT02658435
Title: A Phase 1, Multi-center, Single-masked, Randomized, Placebo-controlled, Parallel-group Study to Investigate the Ophthalmologic Safety and Pharmacodynamics of 300mg Single Doses of Tafenoquine (SB 252263) in Adult Healthy Volunteers
Brief Title: Assessment of Any Potential Retinal Effects of Tafenoquine (TQ)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201807
Record Dates: First submitted 2016-01-04; First posted 2016-01-18 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Malaria, Vivax
Keywords: Malaria; Retinal; Ophthalmic; Plasmodium. vivax; Tafenoquine; Pharmacodynamic
MeSH Terms: conditions — Malaria, Vivax; Malaria | interventions — tafenoquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tafenoquine 300 milligram (mg) single dose (Experimental): Participants will receive single dose of TQ (2 tablets of 150mg) after standard meal. Participant will be randomized in a 2:1 ratio to 300mg TQ (n=300) or matched-placebo (n=150).
  Interventions: Drug: Tafenoquine 150 mg
- Matched Placebo 300mg single dose (Placebo Comparator): Participants will receive single dose of matched placebo (2 tablets of 150mg) after standard meal. Participant will be randomized in a 2:1 ratio to 300mg TQ (n=300) or matched-placebo (n=150).
  Interventions: Drug: Matched placebo 150mg

INTERVENTIONS:
Drug: Tafenoquine 150 mg — Tablet contains TQ as tafenoquine succinate. The 2 tablets (2 tablets of 150mg) of dark pink, capsule-shaped, film coated will be administered orally with 240ml of water.
  Arms: Tafenoquine 300 milligram (mg) single dose
Drug: Matched placebo 150mg — It is the matched Placebo tablet. The 2 tablets (2 tablets of 150mg) of dark pink, capsule-shaped, film coated will be administered orally with 240ml of water.
  Arms: Matched Placebo 300mg single dose

SUMMARY:
The study aims to provide evidence of retinal safety to support the use of tafenoquine as a potential single dose radical cure treatment for patients with Plasmodium vivax (P. vivax) malaria (i.e., co-administration of a schizonticidal drug with TQ). The study will be conducted as a single masked, randomized, placebo-controlled, parallel group design. It will assess retinal changes from baseline using spectral domain optical coherence tomography (OCT) and fundus auto fluorescence (FAF) at Month 3 (90 days) post-dose in adult healthy volunteers (participants). A placebo control group will be used to compare the results in the TQ group. Interim analysis will be conducted after completing 100 out of 300 participants in TQ group and 50 out of 150 participants in matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, brief physical examination, and laboratory tests.
* Participant values for haematology and chemistry within the normal range. A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight between >=35 kilogram (kg) and =<100kg
* Male OR Female. Female participant is eligible to participate if she is not pregnant (as confirmed by a negative [serum or urine, according to site standard] human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as Pre-menopausal females with one of the following: Documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or Hysterectomy or Documented Bilateral Oophorectomy or Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to site specific laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from screening until completion of the Day 90 follow-up visit.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine Aminotransferase (ALT) and bilirubin >1.5 times Upper Limit of Normal (ULN) (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The QT interval corrected (QTc) for heart rate according to Fridericia's formula (QTcF). QTcF > 450 milli second (msec). Other calculation methods (e.g. QT interval corrected for heart rate according to Bazett's formula [QTcB], individually corrected QT interval [QTcI]) machine-read or manually over-read are not acceptable.
* Use of prescription (except female contraception and acetaminophen at doses of =<2 grams(g)/day) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise participant safety.
* History of regular alcohol consumption within 30 days of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Positive results for drugs of abuse
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 30 days prior to screening.
* History of sensitivity to TQ, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* History of thalassaemia; or current or past history of methemoglobinemia or methemoglobin percentage above the reference range at screening.
* Lactating females.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 15 days of dosing with TQ or matched-placebo.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Participants with a hemoglobin values outside the lower limit of normal range. A single repeat is allowed for eligibility determination.
* Documented phenotypic Glucose-6-phosphate dehydrogenase (G6PD) deficiency, determined by a quantitative assay of enzyme activity. Defined as <70% of locally defined median.
* A BCVA (bilateral) at screening of =<72 letters
* Eye disease that could compromise assessment of BCVA or imaging of the posterior pole by fundus photography, or spectral domain OCT, FAF, or is likely to require intervention during the 4 month (approximately) study participation (e.g. cataract, glaucoma with documented visual field loss, ischemic optic neuropathy, retinitis pigmentosa)
* History of retinal vascular disease, retinal detachment, inflammatory disease, central serous chorioretinopathy, or other retinal disease that may affect posterior retinal function or architecture.
* Vitreo-retinal interface disorders (e.g. epiretinal membrane, vitreo-macular traction) that may affect posterior retinal function or architecture
* Intraocular surgery within 3 months of dosing
* Laser photocoagulation within 3 months of dosing
* High Myopia (defined as equal to, or worse than, -6.00 diopters)
* Anterior, intermediate or posterior uveitis (active or history of) or history of significant intraocular infectious disease (e.g., conjunctivitis is not acceptable to include) or another active inflammatory disease
* An OCT central subfield thickness <250 microns or >290 microns
* Presence of significant abnormal patterns on FAF or ocular abnormalities on fundus photography at screening.
* Uncontrolled intraocular pressure >22millimetre of mercury (mmHg).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 486 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Proportion of participants in the TQ group having retinal changes from Baseline in Central subfield thickness and Central retinal lesion thickness | Baseline and Day 90(follow-up)
  The change from baseline will be assessed as a binomial output as, Yes or No. Spectral domain OCT (SD-OCT) images/scan will be obtained. For Central subfield thickness and Central retinal lesion thickness, change from baseline of at least 40 microns (µ) will be consider 'Yes'. Central Retinal Lesion Thickness is defined as the distance between the inner limiting membrane of the retina and the inner border of the choriocapillaris measured in the central 1millimeter (mm) of the centre scan
Proportion of participants in the TQ group having retinal changes from Baseline in Total macular volume | Baseline and Day 90(follow-up)
  The change from baseline will be assessed as a binomial output as, Yes or No. SD-OCT images/scan will be obtained. Total Macular Volume, change from baseline of 10% will be considered 'Yes'
Proportion of participants in the TQ group having retinal changes from Baseline in Ellipsoid zone disruption | Baseline and Day 90(follow-up)
  The change from baseline will be assessed as a binomial output as, Yes or No. SD-OCT images/scan will be obtained. Ellipsoid zone disruption will be assessed by manual reading
Proportion of participants in the TQ group having retinal changes from Baseline in abnormal auto-fluorescence patterns | Baseline and Day 90(follow-up)
  The change from baseline will be assessed as a binomial output as, Yes or No. SD-OCT images/scan will be obtained. Abnormal auto-fluorescence will be assessed by FAF by manual reading

SECONDARY OUTCOMES:
Mean change from baseline in OCT parameter like central retinal thickness as a safety measure | Baseline and Day 90(follow-up)
  SD-OCT images/scan will be obtained. Central retinal thickness is the thickness at the centre point of the macula
Mean change from baseline in OCT parameter like central subfield thickness as a safety measure. | Baseline and Day 90(follow-up)
  SD-OCT images/scan will be obtained. Central subfield thickness measures thickness from top of Internal limiting membrane (ILM) to bottom of Retinal pigment epithelium (RPE).
Mean change from baseline in OCT parameter like central retinal lesion thickness as a safety measure. | Baseline and Day 90(follow-up)
  SD-OCT images/scan will be obtained. Central retinal lesion thickness measures a greatest linear thickness from ILM to inner border of choriocapillaris
Mean change from baseline in OCT parameters;. Total macular volume as a safety measure. | Baseline and Day 90(follow-up)
  SD-OCT images/scan will be obtained. Total macular volume describes the overall thickness of retina from top of ILM to bottom of RPE as a volume measurement.
Mean change from baseline in OCT parameters ;. Ellipsoid zone disruption as a safety measure. | Baseline and Day 90(follow-up)
  SD-OCT images/scan will be obtained. Ellipsoid zone disruption will measure zones of absent or irregular ellipsoid layer.
Changes from baseline in the status of the outer retina/photoreceptor complex as a safety measure. | Baseline and Day 90(follow-up)
  SD-OCT images/scan will be obtained.
Proportion of participants with abnormal changes from baseline observed on FAF as a safety measure. | Baseline and Day 90(follow-up)
  FAF images will be obtained. Qualitative assessment will be done to check for any abnormal patterns of auto-fluorescence in the macular region that may be indicative of disease of the retinal pigment epithelium.
Mean change from baseline in best corrected visual acuity (BCVA) as a safety measure of TQ in comparison to placebo. | Baseline and Day 90(follow-up)
  BCVA will be measured by a trained examiner
Proportion of participants with vortex keratopathy from the slit lamp examination as a safety measure of TQ in comparison to placebo. | Baseline and Day 90(follow-up)
  Vortex keratopathy (corneal deposits) will be confirmed by slit lamp examination. Anterior and posterior segment evaluation will be done.
Number of participants with of adverse events as a safety measure | 90 days
  An AE is any untoward medical occurrence in a participant or clinical investigation temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Baltimore, Maryland

REFERENCES:
- [Derived] Ackert J, Mohamed K, Slakter JS, El-Harazi S, Berni A, Gevorkyan H, Hardaker E, Hussaini A, Jones SW, Koh GCKW, Patel J, Rasmussen S, Kelly DS, Baranano DE, Thompson JT, Warren KA, Sergott RC, Tonkyn J, Wolstenholme A, Coleman H, Yuan A, Duparc S, Green JA. Randomized Placebo-Controlled Trial Evaluating the Ophthalmic Safety of Single-Dose Tafenoquine in Healthy Volunteers. Drug Saf. 2019 Sep;42(9):1103-1114. doi: 10.1007/s40264-019-00839-w. PMID 31187437